CLINICAL TRIAL: NCT05093452
Title: Motivational Interviewing of Parents in Maternity Wards About Vaccination (Entretien Motivationnel Sur la Vaccination auprès Des Parents Dans Les maternités)
Brief Title: MOTIVAC-MATER-Confiance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Observatoire Regional de la Sante Provence-Alpes-Côte d'Azur (Other)
Collaborators: CRES PACA Marseille (Unknown); Institut de Recherche en Santé Publique, France (Other); Hospital St. Joseph, Marseille, France (Other); Hôpital Sainte-Musse CH Toulon (Unknown); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Pierre Verger, Head of ORS PACA (Observatoire Régional de la Santé - Provence-Alpes-Côte-d'Azur), Observatoire Regional de la Sante Provence-Alpes-Côte d'Azur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-01-07-04
Record Dates: First submitted 2021-09-24; First posted 2021-10-26 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Vaccination Promotion
Keywords: Vaccine hesitancy; Motivational interviewing; Childhood vaccination
MeSH Terms: conditions — Vaccination Hesitancy | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Educational session based on the motivational interviewing
  Interventions: Behavioral: Motivational Interviewing
- Information flyer (Other): Information flyer on childhood vaccines
  Interventions: Other: Information flyer

INTERVENTIONS:
Behavioral: Motivational Interviewing — Mothers randomized in the intervention group will receive an educational session based on the motivational interviewing (MI) approach with a midwife. The midwife will have first received a standardized 3 days training session on the content and techniques of MI. The MI intervention will be carried out in simple and understandable language in order to allow discussion and questions from parents rather than provide prescriptive and direct information. The intervention will last approximatively 15 to 20 minutes.
  Arms: Motivational interviewing
Other: Information flyer — Mothers randomized in the control group will receive a locally information flyer on childhood vaccines without any oral explanation by the midwife.
  Arms: Information flyer

SUMMARY:
CONTEXT Vaccination has reduced mortality and morbidity by controlling many vaccine-preventable diseases. To prevent recurrence of these diseases, high vaccine coverages (VCs) (≥ 95%) are needed. But VCs for infants remain suboptimal, and four out of 10 parents doubt the safety and efficacy of vaccines in France. The Ministry of Health therefore decided in July 2017 to expand vaccination requirements to 11 valences now required to enter in young children collective structures. This measure, which went into effect in January 2018, has produced significant effects on VCs, but despite this, vaccine hesitancy (VH) persists in the general population at a prevalence level that fluctuates around 20% to 25%.

Motivational interviewing is a collaborative conversational style that reinforces a person's own motivation and commitment to behavior change. It has been successfully tested in multiple domains related to health behavior change. It has also been adapted in Quebec in the area of vaccination and tested in maternity wards with postpartum mothers (Promovac study). Having led to an increase in the VCs of infants by an average of 7 percentage points and a 40% decrease in vaccine hesitancy, this approach has been in the process of being generalized to all maternity units in Quebec since 2017 (EMMIE program). It is indeed proving to be one of the most effective at present in improving confidence in early childhood vaccines.

OBJECTIVES The main objective of this research is to provide proof of concept that, in the French context of mandatory vaccination for infants but also of high rates of VH, an educational strategy based on the principles and techniques of motivational interviewing and carried out with parents in the maternity ward in the days following delivery can reduce vaccine hesitancy (VH).

The secondary objectives are as follows:

* to verify that this reduction in VH is associated with a change in knowledge, attitudes, and beliefs regarding vaccines;
* to verify that this reduction is sustainable (at 12 months);
* to evaluate the acceptability and satisfaction of the interview for the parents

METHODS This is a pragmatic randomized controlled multicenter study with individual randomization unit comparing the impact of motivational interviewing to a standard care with a leaflet on vaccination.

Motivational interviewing will be carried out by trained midwives from the two participating maternity units (one in Marseille (Bouches-du-Rhône) and the other in Toulon (Var)), as part of the routine care provided to parturients. The midwives will be trained by the founding specialist of motivational interviewing in Quebec, during a two and a half day training course. This training will include a presentation of the theoretical foundations of this approach, its adaptation to the field of vaccination, and interactive games to put it into practice. The trained midwives will then be able to put this approach into practice during a one-month pilot period with parturients, during which they will be able to benefit from support in the form of a debriefing. The actual survey will only start at the end of this pilot phase.

In each group, a questionnaire will be offered to the women (couples) who have agreed to participate, both before the motivational interview (or delivery of the leaflet) and after the interview (or delivery of the leaflet). The second questionnaire will be completed before discharge from the maternity hospital. A third evaluation time is planned at 12 months in both groups: it will be carried out by internet or telephone.

The primary endpoint will be the change in the vaccine hesitancy score, measured by an international scale validated in French (Opel scale).

Secondary endpoints will be changes in knowledge, attitudes and beliefs about vaccination between the two groups as well as satisfaction with the ME and the brochure.

Randomization will be performed in blocks of 8, prior to acceptance for participation in this research.

EXPECTED BENEFITS If the results of this research provide proof of concept that the educational strategy based on motivational interviewing adapted to the vaccination of infants after delivery, in maternity wards, makes it possible, in the French context, to reduce VH, this will be a major advance in public health in France. Indeed, even if the vaccination obligations introduced in January 2018 have had a positive impact on infant vaccination coverage, VH remains present in parents in a proportion that remains worrying (20 to 25% according to surveys). The results of this research will then allow us to study the conditions for generalizing motivational interviewing in order to reinforce confidence in vaccination, which is lacking in a significant part of the French population.

ELIGIBILITY:
Inclusion Criteria:

* Mothers aged 18 years or more
* Mothers residing in the PACA region (Provence-Alpes-Côtes-d'Azur) at the time of the delivery
* Mothers who can read and speak French
* Mothers able to give a free and informed consent
* Mothers who provide written consent

Exclusion Criteria:

* Mothers of new-born needing to be transferred in a 3rd level maternity ward (because of severe condition)
* Mothers who will leave early maternity ward (<24h)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Vaccine hesitancy score (Opel score) | During the 72-hour postpartum stay at the maternity ward
  Parents' vaccine hesitancy score, regarding vaccination of their child, assessed by a questionnaire before and after the intervention at the maternity ward. Using the Opel score (Opel. Validity and reliability of a survey to identify vaccine-hesitant parents. Vaccine. 2011)
Knowledge, attitudes, and beliefs regarding vaccines | During the 72-hour postpartum stay at the maternity ward
  Parents' knowledge, attitudes, and beliefs regarding vaccines, assessed by a questionnaire before and after the intervention at the maternity ward. Using the PromovaQ questionnaire, which was constructed and developed using a composite model inspired by the Health Belief Model and the Theory of Planned Behavior.
  * Dubé. Overview of knowledge, attitudes, beliefs, vaccine hesitancy and vaccine acceptance among mothers of infants in Quebec, Canada. Human Vaccines & Immunotherapeutics. 2018.
  * Gagneur. Promoting vaccination in maternity wards - motivational interview technique reduces hesitancy and enhances intention to vaccinate, results from a multicentre non-controlled pre- and post-intervention RCT-nested study, Quebec, March 2014 to February 2015. Euro Surveillance. 2019.
  * Gagneur. Promoting vaccination in the province of Québec, the PromoVaQ randomized controlled trial protocol. BMC Public Health. 2019.)
Vaccine hesitancy score (Opel score) (sustainability) | 12 months after the intervention at the maternity ward
  Parents' vaccine hesitancy score, regarding vaccination of their child, assessed at 12 months by an online or by-phone questionnaire.
Acceptability and satisfaction of the interview for the parents | During the 72-hour postpartum stay at the maternity ward
  Parents' acceptability and satisfaction of the interview assessed by a questionnaire after the intervention (MI or leaflet) at the maternity ward.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Verger, MD, Principal Investigator — ORS PACA
Locations (2):
- France (2):
  - Hôpital Saint-Joseph, Marseille
  - Hôpital Sainte-Musse, Toulon

IPD SHARING:
Plan to Share IPD: No